CLINICAL TRIAL: NCT02815839
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, Food Effect, Pharmacokinetics, and Pharmacodynamics of Single Doses of SHR4640 in Healthy Subjects
Brief Title: Single Dose Study of SHR4640 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR4640-101
Record Dates: First submitted 2016-04-27; First posted 2016-06-28 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-06

CONDITIONS: Gout; Hyperuricemia
Keywords: urate transporter 1; SHR4640; single ascending dose; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — ruzinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Cohort 1 (Experimental): 2.5-mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: Placebo
- Cohort 2 (Experimental): 5-mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: Placebo
- Cohort 3 (Experimental): 7.5-mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: Placebo
- Cohort 4 (Experimental): 10-mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: Placebo
- Cohort 5 (Experimental): 20-mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: Placebo

INTERVENTIONS:
Drug: SHR4640
Drug: Placebo

SUMMARY:
The objective of the study is to assess the safety, tolerance, food effect, pharmacokinetic and pharmacodynamic properties of single dose adminstration of SHR4640 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body weight≥50, BMI:19-24kg/m2;
* Screening serum urate level ≤ 4.5 mg/dL for male and ≤ 3.5 mg/dL for female;
* Medically stable based on physical examination, medical history, laboratory results, vital sign measurements, and 12-lead electrocardiogram (ECG) at screening;

Exclusion Criteria:

* History of hyperuricemia or gout.
* Pregnancy or breastfeeding;
* History or suspicion of kidney stones;
* serum creatinine>1.5mg/dl for male, >1.2mg/dl for female;
* alanine aminotransferase and/or aspartate aminotransferase>2 upper limit of normal, or total bilirubin>2.5 upper limit of normal.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | Clinical significant changes from baseline up to to Day 15; from baseline up to Day 19 for 7.5mg dose group

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to day 4; up to day 11 for 7.5mg dose group
Area under the plasma concentration versus time curve (AUC) | up to day 4; up to day 11 for 7.5mg dose group
Half-time (T1/2) | up to day 4; up to day 11 for 7.5mg dose group
Time to the peak plasma concentration (Tmax) | up to day 4; up to day 11 for 7.5mg dose group
Cmax of SHR4640 dosed after high-fat meal in 7.5mg dose group | up to day 11
AUC of SHR4640 dosed after high-fat meal in 7.5mg dose group | up to day 11
T1/2 of SHR4640 dosed after high-fat meal in 7.5mg dose group | up to day 11
Tmax of SHR4640 dosed after high-fat meal in 7.5mg dose group | up to day 11
Changes in serum uric acid concentration from baseline | up to day 4; up to day 11 for 7.5mg dose group
  absolute and percent changes in serum acid concentration
Changes in urinary uric acid excretion from baseline | up to day 4; up to day 11 for 7.5mg dose group
  percent changes in urinary uric acid excretion from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Sichuan, China